CLINICAL TRIAL: NCT07206264
Title: Chemotherapy Combined With Targeted Therapy as First-line Treatment for Mantle Cell Lymphoma Based on MRD and PET-CT Assessment: a Multi-center, Phase II Study
Brief Title: Chemotherapy Combined With Targeted Therapy as First-line Treatment for Mantle Cell Lymphoma Based on MRD and PET-CT Assessment
Acronym: ADAPT-MCL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Huilai Zhang, Hulailai Zhang, Tianjin Medical University Cancer Institute and Hospital, Study director, Tianjin Medical University Cancer Institute and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADAPT-MCL
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Mantle Cell Lymphoma
Keywords: Lymphoma; Mantle cell lymphoma; Bendamustine; anti-CD20 monoclonal antibody; Orelabrutinib
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma | interventions — Bendamustine Hydrochloride; orelabrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mantle cell lymphoma: bendamustine + anti-CD20 monoclonal antibody/orelabrutinib + anti-CD20 monoclo (Experimental): Drug: bendamustine + anti-CD20 monoclonal antibody/orelabrutinib + anti-CD20 monoclonal antibody
  Interventions: Drug: Bendamustine + anti-CD20 monoclonal antibody/orelabrutinib + anti-CD20 monoclonal antibody

INTERVENTIONS:
Drug: Bendamustine + anti-CD20 monoclonal antibody/orelabrutinib + anti-CD20 monoclonal antibody — Induction phase (cycle 1-6):
  Bendamustine (90 mg/m², day 1-2) +anti-CD20 monoclonal antibody (375 mg/m², day 0) from cycles 1-4. Patients who achieve CR and MRD negative continue to receive bendamustine (90 mg/m², day 1-2) + anti-CD20 monoclonal antibody (375 mg/m², day 0) from cycles 5-6; MRD positive patients receive orelabrutinib (150 mg) + anti-CD20 monoclonal antibody (375 mg/m², day 0).
  Maintenance phase (cycle 7-24):
  Patients who achieve CR and are MRD negative at cycle 4 receive bendamustine (90 mg/m², day 1-2) + anti-CD20 monoclonal antibody (375 mg/m², day 0); MRD-positive patients receive orelabrutinib (150 mg) + anti-CD20 monoclonal antibody (375 mg/m², day 0).
  Other Names: BR/OR

SUMMARY:
This is a single-arm, multi-center, prospective, phase II study. The primary objective is to assess the efficacy and safety of bendamustine/orelabrutinib combined with an anti-CD20 monoclonal antibody in treatment-naïve patients with mantle cell lymphoma.

DETAILED DESCRIPTION:
Mantle cell lymphoma (MCL) is a subtype of B-cell non-Hodgkin's lymphoma and is considered to be incurable. MCL patients have varied clinical presentations (generally symptomatic to an asymptomatic indolent clinical course). Over the past decade, significant advances in the treatment of MCL have been achieved through intensive immunochemotherapy regimens and clinical trials evaluating novel targeted agents and combination strategies. However, early disease relapse remains a frequent clinical challenge. Recently, combination regimens involving chemotherapy and targeted therapy have demonstrated promising efficacy with acceptable safety profiles. Bendamustine is a unique cytotoxic agent that induces apoptosis through activation of DNA damage stress responses, disruption of mitotic checkpoints, and induction of mitotic catastrophe. Zuberitamab is a novel anti-CD20 monoclonal antibody that demonstrates enhanced antibody-dependent cellular cytotoxicity compared with rituximab. Orelabrutinib is a potent, irreversible, and highly selective Bruton tyrosine kinase inhibitor.

This study is a multicenter, prospective trial involving previously untreated patients with MCL. During the induction phase (cycles 1-4), all patients will receive bendamustine at a dose of 90 mg/m² in combination with anti-CD20 monoclonal antibody at 375 mg/m². After cycle 4, patients who achieve a complete response (CR) and are minimal residual disease (MRD) negative will continue to receive the same regimen (bendamustine 90 mg/m² plus anti-CD20 monoclonal antibody 375mg/m²) for cycles 5 to 6. In contrast, patients who are MRD positive will switch to a treatment regimen consisting of orelabrutinib at 150 mg combined with anti-CD20 monoclonal antibody at 375 mg/m². During the maintenance phase (cycles 7-24), patients who achieve CR and are MRD negative at cycle 4 will continue receiving bendamustine plus anti-CD20 monoclonal antibody, while MRD-positive patients will continue treatment with orelabrutinib plus anti-CD20 monoclonal antibody until disease progression, relapse, intolerable toxicities, death, loss to follow-up, or withdrawal of consent, whichever occurs first, with a maximum of 24 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Gender not limited, aged ≥65 years, or aged ≥60 years but <65 years and unsuitable or unwilling to undergo stem cell transplantation due to the following reasons:

   1. Creatinine clearance rate >30 mL/min, but <70 mL/min;
   2. Presence of other comorbidities that contraindicate high-intensity induction chemotherapy;
   3. High-risk patients who are expected to fail stem cell mobilization and collection (such as those with bone marrow infiltration, diabetes, thrombocytopenia). Patients who are unwilling to receive autologous stem cell transplantation, considering potential complications post-transplantation (such as prolonged bleeding, immunodeficiency, hemorrhage, severe infections), and relapse.
2. Histologically confirmed mantle cell lymphoma at stages II-IV;
3. Patients who have not received prior treatment;
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2;
5. Adequate organ function:

   1. Hematological: Absolute neutrophil count ≥1.5×109/L, platelets ≥75×109/L, hemoglobin ≥75 g/L. If accompanied by bone marrow involvement: Absolute neutrophil count ≥1.0×109/L, platelets ≥50×109/L, hemoglobin ≥50 g/L.
   2. Biochemical: Total bilirubin ≤1.5 times the upper limit of normal (ULN), aspartate transaminase (AST) or alanine transaminase (ALT) ≤2 times ULN.
6. Coagulation function: International normalized ratio (INR) ≤1.5 times ULN;
7. Expected survival time ≥12 months;
8. Voluntarily sign a written informed consent form before the trial screening.

Exclusion Criteria:

1. Progression to higher-grade disease or central nervous system involvement;
2. Uncontrolled or significant cardiovascular diseases:

   1. Within 6 months prior to the first administration of the study drug, there was New York Heart Association (NYHA) class II or higher congestive heart failure, unstable angina pectoris, myocardial infarction, or a need for treatment of arrhythmia at the time of screening, with left ventricular ejection fraction (LVEF) < 50%;
   2. Primary cardiomyopathies (such as dilated cardiomyopathy, hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, restrictive cardiomyopathy, and unclassified cardiomyopathy);
   3. A history of clinically significant QTc interval prolongation, or a QTc interval >470 ms for females or >450 ms for males during the screening period;
   4. Participants with symptomatic or medication-requiring coronary artery disease;
   5. Participants with uncontrolled hypertension, defined as systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg despite adequate therapy with three antihypertensive agents (including a diuretic) for at least one month, or requiring four or more antihypertensive agents to achieve control.
3. Participants with active bleeding within 2 months prior to screening, those currently on anticoagulant therapy, or those deemed by the investigator to have a significant risk of bleeding;
4. History of deep vein thrombosis or pulmonary embolism within the past 6 months;
5. Major surgery within 6 weeks prior to screening or minor surgery within 2 weeks prior to screening. Major surgery is defined as any surgical procedure requiring general anesthesia; diagnostic endoscopy is not considered major surgery;
6. Active infection or uncontrolled hepatitis B virus (HBV) infection (HBsAg positive and/or HBcAb positive with detectable HBV DNA), hepatitis C virus (HCV) antibody positive, HIV/AIDS, or other severe infectious diseases;
7. Participants with pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation-induced lung disease, drug-related lung disease, or other conditions affecting pulmonary function;
8. Pregnant women, breastfeeding women, and fertile participants unwilling to use effective contraception;
9. Participants requiring continuous use of drugs with strong inhibition or induction effects on cytochrome P450 CYP3A4;
10. Other conditions deemed unsuitable for participation in this trial by the investigator.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From the date of the initiation of treatment until the date of first documented progression, up to 2 years.
  PFS is defined as the time from the initiation of treatment to the first occurrence of progression or relapse as assessed by the investigator, or death from any cause. Patients who remain alive and progression-free at the data cutoff date, PFS will be censored at the last tumor assessment date.

SECONDARY OUTCOMES:
Overall response rate (ORR) | From the initiation of treatment to the end of therapy, up to 2 years.
  The ORR is defined as the proportion of patients with a response of CR or PR.
Complete response rate (CRR) | From the initiation of treatment to the end of therapy, up to 2 years.
  Complete response rate is defined as the proportion of patients with a response of CR.
Duration of Response (DOR) | From the first demonstration of response until disease progression/death, up to 2 years.
  DOR is defined as the time from documentation of response to treatment to the first documentation of tumor progression or death due to any cause, whichever comes first.
Time to response (TTR) | From the start of therapy to the first documentation of response.
  TTR is defined as the time from the start of therapy to the first response.
Overall survival (OS) | From the date of the initiation of treatment until the date of death, up to 3 years.
  OS is defined as the time from the initiation of treatment to death from any cause. Patients alive at the data cutoff date will have their OS censored at the date of the last follow-up.
Adverse events (AEs) | From the date of enrollment until the date of death, up to 3 years.
  AEs will be graded according to the NCI-CTCAE Version 5.0.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Hebei Medical University Tumor Hospital, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Shandong Cancer Hospital, Jinan, Shandong
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No